CLINICAL TRIAL: NCT01118910
Title: Open-Label Pilot Study of the Efficacy and Safety of Vusion Ointment for the Treatment of Intertrigo
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Image Dermatology P.C. (Other)
Responsible Party: Jeanine B. Downie, M.D., Image Dermatology P.C.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W0319-501
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Intertrigo
Keywords: Intertrigo; Vusion
MeSH Terms: conditions — Intertrigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vusion ointment (Experimental)
  Interventions: Drug: Vusion

INTERVENTIONS:
Drug: Vusion — Vusion will be applied to areas of intertrigo

SUMMARY:
The purpose of this study is to determine if people with moist, red, patches on their skin in body folds would benefit treatment of those areas with an FDA-approved drug called Vusion.

DETAILED DESCRIPTION:
Intertrigo is an inflammatory condition of skin folds, induced or aggravated by heat, moisture, maceration, friction, or lack of air circulation. It is typically chronic with insidious onset of itching, burning, and stinging within the affected skin folds. Intertrigo frequently worsened or colonized by infection, which most commonly is candidal but also may be bacterial, fungal, or viral. The etiology of diaper dermatitis shows significant overlap with that of intertrigo. Vusion ointment, a highly effective treatment for diaper dermatitis, has been used by physicians for the treatment of intertrigo; however, there is a paucity of data in the literature regarding the use of Vusion ointment in this indication.

This study is the first to formally investigate the efficacy and safety of Vusion ointment for the treatment of intertrigo.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of intertrigo

Exclusion Criteria:

* Pregnancy
* Use of systemic or topical antifungal or corticosteroid treatment in the previous 14 days or during the 3-month treatment period
* allergy of sensitivity to Vusion
* undergoing warfarin anticoagulation
* alcohol or drug abuse
* Investigator determines they cannot particpate
* history of non-compliance or poor cooperation
* participation in an investigaitonal drug study within 30 days of Baseline Visit

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The number of patients for whom Vusion effectively treated intertrigo | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeanine B. Downie, M.D., Principal Investigator — Image Dermatology P.C.
Locations (1):
- Image Dermatology P.C., Montclair, New Jersey, United States